CLINICAL TRIAL: NCT05373212
Title: A Trial Investigating the Dose Linearity and Safety of BC Combo THDB0207 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CT048-ADO05
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Intervention Model Description: Four-period crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BC Combo THDB0207 Low dose (Experimental): Single administration of BC Combo THDB0207 (Low dose)
  Interventions: Drug: Euglycemic clamp with BC Combo THDB0207
- BC Combo THDB0207 Medium dose (Experimental): Single administration of BC Combo THDB0207 (Medium dose)
  Interventions: Drug: Euglycemic clamp with BC Combo THDB0207
- BC Combo THDB0207 High dose (Experimental): Single administration of BC Combo THDB0207 (High dose)
  Interventions: Drug: Euglycemic clamp with BC Combo THDB0207
- Humalog® Mix25 (Active Comparator): Single administration of Humalog® Mix25
  Interventions: Drug: Euglycemic clamp with Humalog® Mix25

INTERVENTIONS:
Drug: Euglycemic clamp with BC Combo THDB0207 — Administration of a single dose of BC Combo THDB0207 during an euglycemic clamp procedure.
  Arms: BC Combo THDB0207 High dose; BC Combo THDB0207 Low dose; BC Combo THDB0207 Medium dose
Drug: Euglycemic clamp with Humalog® Mix25 — Administration of a single dose of Humalog® Mix25 during an euglycemic clamp procedure.
  Arms: Humalog® Mix25

SUMMARY:
This is a randomised, double-blind, four-period crossover euglycaemic clamp trial in subjects with type 2 diabetes.

Each subject will be randomly allocated to one of four treatment sequences. Each sequence will comprise 3 different single doses of BC Combo THDB0207 (Low dose, Medium dose, and High dose) and one single dose of Humalog® Mix25.

Subjects will come to the clinical trial centre in a fasted state in the morning of each dosing day and stay at the clinical trial centre until the 30-hour clamp procedures have been terminated.

DETAILED DESCRIPTION:
Subjects will attend the study site in the morning in a fasted state and will be connected to an automated glucose clamp device. Prior to dose administration plasma glucose will be stabilised at a target level of 100 mg/dL by means of an intravenous infusion of glucose or insulin. IMP administration will be done by an unblinded person by means of subcutaneous injections in the abdominal wall.

Following each dosing a euglycaemic glucose clamp procedure will be carried out for up to 30 hours.

The pharmacodynamic assessment will be based on the time course of glucose infusion rate (GIR) and plasma glucose.

Plasma insulin concentrations will be measured using a specific validated bioanalytical method differentiating concentrations of insulin glargine, of its main metabolites insulin-glargine-M1 and insulin-glargine-M2, and of insulin lispro. Pharmacokinetic assessments will be based on total insulin concentration (insulin glargine + insulin glargine-M1 + insulin glargine-M2 + insulin lispro), on insulin glargine concentration (insulin glargine + insulin glargine-M1 + insulin glargine-M2), or on insulin lispro concentration.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (as diagnosed clinically) for ≥ 12 months
* HbA1c ≤9.0%
* Total insulin dose of < 1.2 U/kg/day
* Body mass index between 20.0 and 35.0 kg/m2 (both inclusive)
* Treated with a stable insulin regimen for ≥ 3 months prior to screening

Exclusion Criteria:

* Known or suspected hypersensitivity to the IMPs or any of the excipients or to any component of the IMP formulation
* Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomisation in this trial
* Clinically significant abnormal screening laboratory tests, as judged by the Investigator considering the underlying disease
* Clinically relevant comorbidity, capable of constituting a risk for the subject when participating in the trial or of interfering with the interpretation of data
* Systolic blood pressure < 90 mmHg or >160 mmHg and/or diastolic blood pressure < 50 mmHg or > 95 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension)
* Heart rate at rest outside the range of 50-90 beats per minute
* Use of GLP-1 receptor agonists or oral antidiabetic drugs (OADs) other than stable intake of metformin within 4 weeks prior to screening
* Women of childbearing potential who are not using a highly effective contraceptive method

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
AUCTOTAL0-last | From t=0 to t=30 hours after IMP administration
  Area under the total insulin concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
CmaxTOTAL | From t=0 to t=30 hours after IMP administration
  Maximum total insulin concentration

SECONDARY OUTCOMES:
AUCGIR 0-last | From t=0 to t=30 hours after IMP administration
  Area under the glucose infusion rate curve from 0 hours until the end of clamp
GIRmax | From t=0 to t=30 hours after IMP administration
  Maximum glucose infusion rate
tGIRmax | From t=0 to t=30 hours after IMP administration
  Time to maximum glucose infusion rate
Tonset of action | From t=0 to t=30 hours after IMP administration
  Time until Plasma Glucose (PG) has decreased by at least 5 mg/dL from the baseline PG value.
AUCGIR 0-6h | From t=0 to t=6 hours
  Area under the glucose infusion rate curve from t=0 hours to t=6 hours
AUCTOTALlast | From t=0 to t=30 hours after IMP administration
  Area under the insulin concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
AUCTOTAL 0-1h | From t=0 to t=1 hour
  Area under the total insulin concentration-time curve from t=0 to t=1 hour
AUCTOTAL 0-2h | From t=0 to t=2 hours
  Area under the total insulin concentration-time curve from t=0 to t=2 hours
AUCTOTAL 0-6h | From t=0 to t=6 hours
  Area under the total insulin concentration-time curve from t=0 to t=6 hours
AUCTOTAL 2-6h | From t=2 to t=6 hours
  Area under the total insulin concentration-time curve from t=2 to t=6 hours
AUCTOTAL 6-12h | From t=6 to t=12 hours
  Area under the total insulin concentration-time curve from t=6 to t=12 hours
AUCTOTAL 6-24h | From t=6 to t=24 hours
  Area under the total insulin concentration-time curve from t=6 to t=24 hours
AUCTOTAL 12-24h | From t=12 to t=24 hours
  Area under the total insulin concentration-time curve from t=12 to t=24 hours
AUCTOTAL 12-30h | From t=12 to t=30 hours
  Area under the total insulin concentration-time curve from t=12 to t=30 hours
AUCTOTAL 0-30h | From t=0 to t=30 hours
  Area under the total insulin concentration-time curve from t=0 to t=30 hours
CTOTALmax | From t=0 to t=30 hours after IMP administration
  Maximum insulin concentration
tmaxTOTAL | From t=0 to t=30 hours after IMP administration
  Time to maximum total insulin concentration
AUCGLA 0-last | From t=0 to t=30 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
AUCGLA 0-1h | From t=0 to t=1 hour after IMP administration
  Area under the insulin glargine concentration-time curve from t=0 to t=1 hour
AUCGLA 0-2h | From t=0 to t=2 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=0 to t=2 hours
AUCGLA 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=0 to t=6 hours
AUCGLA 2-6h | From t=2 to t=6 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=2 to t=6 hours
AUCGLA 6-12h | From t=6 to t=12 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=6 to t=12 hours
AUCGLA 12-24h | From t=12 to t=24 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=12 to t=24 hours
AUCGLA 12-30h | From t=12 to t=30 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=12 to t=30 hours
AUCGLA 0-30h | From t=0 to t=30 hours after IMP administration
  Area under the insulin glargine concentration-time curve from t=0 to t=30 hours
CmaxGLA | From t=0 to t=30 hours after IMP administration
  Maximum concentration of insulin glargine
tmaxGLA | From t=0 to t=30 hours after IMP administration
  Time to maximum insulin glargine concentration
AUCLIS0-last | From t=0 to t=30 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
AUCLIS 0-1h | From t=0 to t=1 hour after IMP administration
  Area under the insulin lispro concentration-time curve from t=0 to t=1 hour
AUCLIS 0-2h | From t=0 to t=2 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=0 to t=2 hours
AUCLIS 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=0 to t=6 hours
AUCLIS 2-6h | From t=2 to t=6 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=2 to t=6 hours
AUCLIS 6-12h | From t=6 to t=12 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=6 to t=12 hours
AUCLIS 12-24h | From t=12 to t=24 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=12 to t=24 hours
AUCLIS 12-30h | From t=12 to t=30 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=12 to t=30 hours
AUCLIS 0-30h | From t=0 to t=30 hours after IMP administration
  Area under the insulin lispro concentration-time curve from t=0 to t=30 hours
CmaxLIS | From t=0 to t=30 hours after IMP administration
  Maximum concentration of insulin lispro
tmaxLIS | From t=0 to t=30 hours after IMP administration
  Time to maximum insulin lispro concentration
Adverse Events | From the first IMP administration to the follow-up visit (i.e. up to 14 weeks)
  Incidence of Adverse Events
Local tolerability | From the first IMP administration to the follow-up visit (i.e. up to 14 weeks)
  Incidence of Injection Site Reactions

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany